CLINICAL TRIAL: NCT00596232
Title: Investigating Mucinase Activity in Airway Disease
Acronym: Mucinase
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-05418; 5P01HL107202-03 (NIH)
Record Dates: First submitted 2008-01-02; First posted 2008-01-16 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Asthma; Cystic Fibrosis
MeSH Terms: conditions — Asthma; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Asthma: People who have been diagnosed with Asthma
- Cystic Fibrosis: People who have been diagnosed with Cystic Fibrosis
- Healthy: People who are non-asthmatic, non smokers with less than 10 pack years and who do not have cystic fibrosis

SUMMARY:
The purpose of this study is to investigate how mucus (phlegm or spit) is broken down once it forms in the airways (bronchial tubes) of people with lung disease. This research study will also examine whether blood groups have an effect on lung function or the type of mucus found in the lung. This study is not designed to be a treatment for asthma, emphysema, cystic fibrosis, or other lung disease. It is designed to help the investigators learn more about the causes of airway disease.

DETAILED DESCRIPTION:
Accumulation of mucus in the airway involves the process of overproduction and reduced clearance of mucin glycoproteins. To date, little attention has been focused on mechanisms of mucin clearance from the airway. We hypothesize that there is enzymatic degradation of mucins ("mucinase activity") in the airway, which acts to break down mucins and facilitate their clearance. We further hypothesize that glycosidases function as mucinases by removing peripheral monosaccharides from oligosaccharides, including oligosaccharides on mucins. Removal of terminal or capping sugars on mucin side chains may be an important mechanism in mucin degradation and clearance from the lung. If mucinase activity exists in the airway then mucus collected from human subjects should demonstrate evidence of mucin degradation ex vivo, especially at 37º celsius. As part of our protocol we propose to examine changes in airway mucus ex vivo under different experimental conditions. Our primary readout will be measures of sputum rheology, namely viscosity and elasticity. Our consultant for this methodology will be Dr Susan Muller (Chemical Engineering, University of California, Berkeley). In order to conduct experimental studies in this way we will need multiple samples from the same subjects. Thus, up to 10 or more sputum samples per subject will be collected on different days. In addition, we are interested in the biochemical properties of sputum and saliva, specifically the composition of mucin molecules found in these fluids.

ELIGIBILITY:
Inclusion Criteria:

Asthma:

1. Male and female subjects aged 18 - 70 years
2. Medical history consistent with asthma
3. PC20 (provocative concentration causing a 20% fall) methacholine ≤ 8 mg/ml for subjects not taking inhaled corticosteroids
4. PC20 methacholine ≤ 16 mg/ml for subjects taking inhaled corticosteroids
5. Ability to provide informed consent

Cystic Fibrosis:

1. Male and female subjects aged 18-55 years
2. Prior diagnosis of cystic fibrosis
3. Ability to provide informed consent

Healthy:

1. Male and female subjects aged 18-70 years
2. No current smoking history
3. No history of asthma or allergic rhinitis
4. FEV1 (forced expiratory volume in 1 second) > 80% predicted
5. Ability to provide informed consent

Exclusion Criteria:

1. Recent heart attack or stroke
2. Known aortic or cerebral aneurysm
3. Uncontrolled hypertension
4. Pregnancy
5. Lactation
6. Lung disease other than asthma,cystic fibrosis, or chronic obstructive pulmonary disease (COPD)/emphysema/chronic bronchitis
7. Upper- or lower-respiratory tract infection 6 weeks prior to study enrollment
8. Significant asthma exacerbation 6 weeks prior to study enrollment
9. Increasing hyposensitization therapy for the past 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers are recruited from community advertisements and health clinics
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2003-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
rheological measurements (viscosity and elasticity) in sputum. | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, M.D., M.Sc., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu